CLINICAL TRIAL: NCT05999799
Title: A Phase 2b, Randomized, Double-Blind, Parallel Group, Placebo Controlled, Dose Finding Study to Evaluate the Efficacy, Safety, Pharmacokinetics, and Pharmacodynamics of GSK1070806 SC Injection in Adult Participants With Moderate to Severe Atopic Dermatitis
Brief Title: A Dose Finding Study to Investigate the Safety and Effectiveness of GSK1070806 in Adult Participants With Moderate to Severe Atopic Dermatitis
Acronym: AtDventure
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision to early terminate the study based on the pre-defined futility criterion for efficacy. No safety concerns were identified.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 219538; 2023-505414-15-00 (Registry Identifier: CTIS)
Record Dates: First submitted 2023-08-11; First posted 2023-08-21 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Dermatitis, Atopic
Keywords: Dermatitis; Atopic; GSK1070806; 219538; Eczema; Skin Diseases; Safety; Efficacy; Immune System Diseases
MeSH Terms: conditions — Dermatitis, Atopic; Dermatitis; Eczema; Skin Diseases; Immune System Diseases | interventions — GSK1070806

STUDY DESIGN:
Intervention Model Description: This is a dose finding, placebo-controlled study where participants will be randomized to receive either GSK1070806 or placebo.
Who Masked: Participant, Investigator
Masking Description: Participants and investigator are blinded to study intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- GSK1070806 Dose 1 (Experimental): Participants will receive GSK1070806 dose 1.
  Interventions: Drug: GSK1070806
- GSK1070806 Dose 2 (Experimental): Participants will receive GSK1070806 dose 2.
  Interventions: Drug: GSK1070806
- GSK1070806 Dose 3 (Experimental): Participants will receive GSK1070806 dose 3.
  Interventions: Drug: GSK1070806
- GSK1070806 Dose 4 (Experimental): Participants will receive GSK1070806 dose 4.
  Interventions: Drug: GSK1070806
- Placebo (Placebo Comparator): Participants will receive placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK1070806 — GSK1070806 will be administered.
  Arms: GSK1070806 Dose 1; GSK1070806 Dose 2; GSK1070806 Dose 3; GSK1070806 Dose 4
Drug: Placebo — Placebo will be administered.
  Arms: Placebo

SUMMARY:
This study is parallel group, placebo-controlled dose-ranging study to evaluate the efficacy, safety, pharmacokinetics, and pharmacodynamics of GSK1070806 in adult participants with moderate to severe Atopic Dermatitis (AtD), who have previously been treated with medicated topical treatments or a biologic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants 18 years to 75 years of age
* Participants with:

  * AtD defined by the AAD Consensus Criteria.
  * Diagnosis of AtD ≥1 year.
  * An IGA score ≥3.
  * AtD involvement of ≥10% body surface area (BSA).
  * EASI score ≥16
  * Baseline pruritus numerical rating scale average score for maximum intensity of at least 3.
* Participants may have had exposure to 1 biologic therapy meeting at least 1 of the following conditions:

  * Participants who stopped treatment due to non-response, partial response, loss of efficacy.
  * Participants who stopped treatment due to intolerance or AEs.
* Participant with a recent history less than or equal to (≤6) months prior to the Screening visit) of inadequate response to a stable regimen of prescription topical medication.
* Participants for whom prescription topical medications are not tolerated.
* Contraceptive use by women should be consistent with local regulations regarding the methods of contraception for those participating in clinical study

Exclusion Criteria:

* Chronic or acute infection requiring treatment with oral or IV antibiotics, antivirals, anti-protozoal, or antifungals within 4 weeks before the Screening visit or anytime between the Screening and Baseline visits.
* Superficial skin infections within 1 week before the Screening visit or active infections (including localized infections), or history of recurrent infections (excluding recurrent fungal infections of the nail bed)
* Known, pre-existing or suspected parasitic infection within 6 months before the Screening visit.
* Symptomatic herpes zoster within 3 months prior to screening
* Uncontrolled hypertension.
* Current or chronic history of liver disease or known hepatic or biliary abnormalities.
* Known or suspected history of immunosuppression, including history of invasive opportunistic infections despite infection resolution or unusually frequent, recurrent, or prolonged infections, per the Investigator's judgment.
* Lymphoma, leukemia, or any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years
* Breast cancer within the past 10 years.
* History or presence of significant medical illness including but not limited to cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematologic, neurological, or psychiatric disorders which in the opinion of the investigator would interfere with the study procedures and/or assessments.
* Previously treated with any oral Janus Kinase inhibitor (JAKi) or other kinase inhibitors, experimental or approved.
* Uncontrolled chronic disease that might require bursts of oral corticosteroids, e.g., co-morbid severe uncontrolled asthma.
* Presence of Hepatitis B surface antibody (HBsAg) or Hepatitis B core antibody (HBcAb) at screening or within 3 months prior to first dose of study intervention.
* Positive hepatitis C antibody test result at screening or within 3 months prior to starting study intervention.
* Positive hepatitis C RNA test result at screening or within 3 months prior to first dose of study intervention.
* Positive HIV antibody test.
* Evidence of active or latent TB as documented by medical history, examination, and TB testing with a positive QuantiFERON test at initial Screening visit.
* Pregnant or breastfeeding women, or women planning to become pregnant or breastfeed during the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2023-11-16 (Actual); Primary Completion 2025-07-23 (Actual); Study Completion 2025-07-23 (Actual)

PRIMARY OUTCOMES:
Percent Change from Baseline (PCFB) in the Eczema Area and Severity Index (EASI) at Week 16 | Baseline and Week 16
  EASI is an internationally used classification for AtD severity and an investigator-assessed measure that is used to assess the extent (area) and severity of AtD. The range of the scale is 0-72, with a higher score indicating greater severity.

SECONDARY OUTCOMES:
Percent Change from Baseline (PCFB) EASI Score for GSK1070806 at Each Time Point | Baseline and up to Week 16
  EASI score percent changes from baseline at each time point will be reported. EASI is an internationally used classification for AtD severity and an investigator-assessed measure that is used to assess the extent (area) and severity of AtD. The range of the scale is 0-72, with a higher score indicating greater severity.
Number of Participants Achieving EASI Reduction of Greater than or Equal to (≥) 75 Percent (%) from Baseline at Week 16 | Baseline and Week 16
  The occurrence of ≥75% reduction from baseline achieving EASI75 score at Week 16 will be reported. EASI is an internationally used classification for AtD severity and an investigator-assessed measure that is used to assess the extent (area) and severity of AtD. The range of the scale is 0-72, with a higher score indicating greater severity.
Number of Participants Achieving Investigator's Global Assessment (IGA) score of 0 or 1 and a Reduction from Baseline ≥ 2 Points at Week 16 | Baseline and up to Week 16
  IGA for AtD is a measure of overall disease severity at the time of assessment on a 5-point scale by the investigator. Where 0-clear, 1-almost clear, 2-mild disease, 3-moderate disease, and 4- severe disease. Higher score indicates severity of disease. A participant with an IGA score of 0 or 1 and a reduction from baseline ≥ 2 points will be reported.
Change from Baseline in Peak Pruritus Numerical Rating Scale (PP-NRS) Score at Week 16 | Baseline and Week 16
  PP-NRS is a patient reported measure of pruritus (itch) intensity assessing worst itch (in the past 24 hours). The values will be evaluated using an 11-point scale (from 0 to 10), with 0 being no itch and 10 being the worst imaginable itch.
Number of Participants Achieving PP-NRS Reduction of ≥4 points from Baseline at Week. 16 | Baseline and Week 16
  Participants achieving a reduction of ≥4 points from baseline of peak pruritus NRS score at Week 16 will be reported. The values will be evaluated using an 11-point scale (from 0 to 10), with 0 being no itch and 10 being the worst imaginable itch.
Number of Participants Achieving EASI Reduction of ≥50%, 90% or 100% from Baseline at Week 16 | Baseline and Week 16
  The occurrence of ≥50%, 90% or 100% reduction from baseline achieving EASI score at Week 16 will be reported. EASI is an internationally used classification for AtD severity and an investigator-assessed measure that is used to assess the extent (area) and severity of AtD. The range of the scale is 0-72, with a higher score indicating greater severity.
Number of Participants Achieving Scoring Atopic Dermatitis (SCORAD) Reduction of ≥ 50% or ≥75% from Baseline at Week 16 | Baseline and Week 16
  Participants achieving a reduction SCORAD reduction of 50% or 75% from Baseline will be reported. SCORAD is a clinical tool to assess the extent and severity of AtD with 3 components. The total score for SCORAD index formula is computed as formula A is defined extent of disease (0-102%), B is defined as the intensity (0-18) and C is defined as the subjective symptoms (0-20). The total SCORAD score ranges from 0 (no disease) to 103 (severe disease).
Change from Baseline in the Body surface area (BSA) of GSK1070806 at Week 16 | Baseline and Week 16
  The BSA assessment estimates the extent of disease or skin involvement with respect to AtD and is expressed as a percentage of total body surface. BSA will be determined by the Investigator or designee using the patient palm = 1% rule
Change from Baseline in the SCORAD of GSK1070806 at Week 16 | Baseline and Week 16
  SCORAD is a clinical tool to assess the extent and severity of AtD with 3 components. The total score for SCORAD index formula is computed as formula A is defined as the extent of disease (0-102%), B is defined as the intensity (0-18) and C is defined as the subjective symptoms (0-20). The total SCORAD score ranges from 0 (no disease) to 103 (severe disease).
Change from Baseline in Patient Reported Outcomes (PRO) Measure of Skin Pain Numerical Rating Scale (SP-NRS) at Week 16 | Baseline and Week 16
  SP-NRS is a patient reported measure assessing worst level of skin pain (in the past 24 hours). The values will be evaluated using an 11-point scale from 0 to 10, with 0 being no pain and 10 being the worst pain imaginable.
Change from Baseline in PRO Measure of Patient Reported Outcomes Measurement Information System (PROMIS) -Sleep Disturbance 8b at Week 16 | Baseline and Week 16
  The PROMIS Short Form Sleep disturbance 8b is a PRO instrument designed to assess self-reported sleep disturbance for which the recall period is the past 7 days. The items are rated on a 5-point verbal rating scale. Items are summed giving a range in raw score from 8 to 40, with higher scores indicating greater severity of sleep disturbance.
Change from Baseline in PRO Measure of Functional Assessment of Chronic Illness Therapy (FACIT) - Fatigue at Week 16 | Baseline and Week 16
  The FACIT-Fatigue scale is a short, 13-item measure that assesses self-reported fatigue and its associated impact for daily activities over the past week. The items are rated on a 5-point Likert-type scale (i.e., 4 = not at all to 0 = very much). The scale range is 0 to 52, with 0 being the worst possible score and 52 indicating no fatigue.
Change from Baseline in PRO Measure of Brief Fatigue Inventory (BFI) - Item 3 at Week 16 | Baseline and Week 16
  The BFI is a self-administered questionnaire developed to assess fatigue severity. The BFI has 9 items. BFI item 3 assesses the worst level of fatigue related concepts (i.e., tiredness, weariness) during the past 24 hours. Participants report their worst level of fatigue daily, for the previous 24 hours, using a numerical rating scale ranging from 0 (no fatigue) to 10 (as bad as you can imagine).
Change from Baseline in PRO Measure of Patient Oriented Eczema Measure (POEM) at Week 16 | Baseline and Week 16
  POEM is a 7-item questionnaire that assesses symptoms of dryness, itching, flaking, cracking, sleep loss, bleeding, and weeping over the last week. The scoring symptom ranges from 0 (absent disease) to 28 (severe disease). Higher score indicates poor QoL.
Change from Baseline in PRO Measure of Dermatology Life Quality Index (DLQI) at Week 16 | Baseline and Week 16
  The DLQI is a 10-item questionnaire that asks participants to evaluate the degree that their skin disease has affected their QoL. It is calculated by summing the scores of the 10 questions, ranging from 0 to 30 with higher scores indicating more impaired QoL. A score of 0 or 1 means that the disease has no effect at all.
Change from Baseline in PRO Measure of Hospital Anxiety and Depression Scale (HADS) at Week 16 | Baseline and Week 16
  The HADS is a self-reported questionnaire which measures depression and generalized anxiety, in the past week. Each item on the questionnaire ranges from 0 (no, not at all) to 3 (yes, definitely). The scale ranges from 0 to 21, with lower score indicating better QoL.
Change from Baseline in PRO Measure of Work Productivity and Activity Impairment Questionnaire-Atopic Dermatitis (WPAI- AD) at Week 16 | Baseline and Week 16
  The WPAI-AD is a validated, patient-reported, quantitative assessment of absenteeism (work time missed), presentism (reduced on-the-job effectiveness), work productivity loss and activity impairment due to a specific health problem.
Occurrences of Adverse Events (AEs), Serious AE (SAEs), and AEs of Special Interest (AESI) | Up to Week 28
  AEs, SAEs, and AESIs will be reported. An AE is any untoward medical occurrence in participant, temporally associated with use of study intervention, whether or not considered related to medicinal product. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect, medically important were categorized as SAE. AESIs of the study drug includes serious and opportunistic infections, serious hypersensitivity reactions and Injection site reactions.
Change from Baseline in Haematology Parameter: Haemoglobin (Hb) (Grams per Litre) | Baseline and Up to Week 28
Change from Baseline in Haematology Parameters: Neutrophils, Lymphocytes, Monocytes, Eosinophils, Basophils, White Blood Cell (WBC), and Platelet Count (Giga Cells per Litre) | Baseline and Up to Week 28
Change from Baseline in Clinical Chemistry Parameters: Alanine Aminotransferase (ALT), Gamma-Glutamyl Transferase (GGT), and Alkaline Phosphatase (AP) (Units per Litre) | Baseline and Up to Week 28
Change From Baseline in Clinical Chemistry Parameters: Aspartate Aminotransferase (AST) (International Units per Litre) | Baseline and Up to Week 28
Change from Baseline in Clinical Chemistry Parameter: Total Bilirubin (Micromoles per Litre) | Baseline and Up to Week 28
Number of Participants with Greater than or Equal to (≥) Grade 3 Hematological/Clinical Chemistry Abnormalities According to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCICTCAE) | Up to Week 28
  Hematological/clinical chemistry abnormalities summarized according to NCI CTCAE grade.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (77):
- United States (16):
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, North Little Rock, Arkansas
  - GSK Investigational Site, Canoga Park, California
  - GSK Investigational Site, Fountain Valley, California
  - GSK Investigational Site, Northridge, California
  - GSK Investigational Site, Oceanside, California
  - GSK Investigational Site, Santa Monica, California
  - GSK Investigational Site, Homestead, Florida
  - GSK Investigational Site, Oakland Park, Florida
  - GSK Investigational Site, Fayetteville, Georgia
  - GSK Investigational Site, Thomasville, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Troy, Michigan
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Dublin, Ohio
  - GSK Investigational Site, West Lake Hills, Texas
- Argentina (6):
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Capital Federal
  - GSK Investigational Site, Ciudad Autonoma de Bueno
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, Mendoza
  - GSK Investigational Site, Rosario
- Bulgaria (2):
  - GSK Investigational Site, Pleven
  - GSK Investigational Site, Sofia
- Canada (5):
  - GSK Investigational Site, Kelowna, British Columbia
  - GSK Investigational Site, Barrie, Ontario
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Markham, Ontario
  - GSK Investigational Site, Québec, Quebec
- China (8):
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Chongqing
  - GSK Investigational Site, Fuzhou
  - GSK Investigational Site, Guangzhou
  - GSK Investigational Site, Hangzhou
  - GSK Investigational Site, Shanghai
  - GSK Investigational Site, Yinchuan
  - GSK Investigational Site, Yiwu
- GSK Investigational Site, Prague, Czechia
- France (2):
  - GSK Investigational Site, La Rochelle
  - GSK Investigational Site, Paris
- Germany (3):
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
  - GSK Investigational Site, Münster
- GSK Investigational Site, Athens, Greece
- Italy (5):
  - GSK Investigational Site, Bari
  - GSK Investigational Site, Bologna
  - GSK Investigational Site, Florence
  - GSK Investigational Site, Modena
  - GSK Investigational Site, Roma
- Japan (7):
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Gunma
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Saitama
- Mexico (4):
  - GSK Investigational Site, Chihuahua City
  - GSK Investigational Site, Durango
  - GSK Investigational Site, Guadalajara
  - GSK Investigational Site, Monterrey
- GSK Investigational Site, Panama City, Panama
- Poland (6):
  - GSK Investigational Site, Chojnice
  - GSK Investigational Site, Elblag
  - GSK Investigational Site, Katowice
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Szczecin
  - GSK Investigational Site, Warsaw
- South Korea (2):
  - GSK Investigational Site, Ansan
  - GSK Investigational Site, Seoul
- Spain (6):
  - GSK Investigational Site, Alicante
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, Granada
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Vigo
  - GSK Investigational Site, Zaragoza
- Thailand (2):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Pathum Thani

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/